CLINICAL TRIAL: NCT01211847
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study Assessing the Efficacy, Safety and Tolerability of Diazoxide Choline Controlled-Release Tablet (DCCR) in Subjects Without Diabetes Mellitus Having Very High Fasting Triglyceride Levels, With Double-Blind DCCR-Fenofibrate Combination Extension
Brief Title: Efficacy Study of Diazoxide Choline to Treat Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Essentialis, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT013
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Hypertriglyceridemia; Dyslipidemia
Keywords: triglycerides; Apo B; non-HDL; statin; fenofibrate
MeSH Terms: conditions — Hypertriglyceridemia; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DCCR (Experimental): DCCR Treatment with 290 mg Diazoxide Choline
  Interventions: Drug: Diazoxide Choline Controlled-Release Tablet
- Placebo (Placebo Comparator): Placebo matching DCCR
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diazoxide Choline Controlled-Release Tablet — DCCR 290 mg once a day for 126 days
  Arms: DCCR
Drug: Placebo — Placebo matching DCCR
  Arms: Placebo

SUMMARY:
Once a day oral administration with DCCR helps lower triglycerides

DETAILED DESCRIPTION:
The population will consist of Statin-naive and Statin-treated subjects, all without diabetes mellitus, with fasting triglyceride levels in the range of ≥ 500 mg/dL and < 1500 mg/dL.

Subjects will be randomly assigned to 1 of 2 treatment groups: DCCR and Placebo

Approximately 44 subjects will be enrolled in the study and stratified by Statin use at a 1:1 ratio in each treatment group,

ELIGIBILITY:
INCLUSION CRITERIA:

Fasting triglycerides

* Difference between Visit 3 (7 days prior to Baseline Visit) and Visit 4 (3 days prior to Baseline Visit) ≤ 60% (compared to the higher value of Visit 3 or Visit 4)
* Run-in Triglycerides* ≥ 500 mg/dL and < 1500 mg/dL *Run-in Triglyceride is defined as the average fasting triglycerides for Visit 3 (7 days prior to Baseline Visit) and Visit 4 (3 days prior to Baseline Visit).

Statin use • Either Statin-naive

* Must not be on statin at Screening and remaining as such during the Run-in/Washout Period and throughout the study

  • Or Statin-treated
* Must be on Lipitor 20 mg initiated at the start of the Run-in/Washout Period and continue throughout the study

Medication washout

* All subjects must be willing to undergo washout of all other lipid-lowering medications

Glycemic status

* Fasting glucose < 126 mg/dL at Screening Visit
* HbA1c < 6.5% at Screening Visit

EXCLUSION CRITERIA:

Medications: recent, current, anticipated

* Administration of investigational drugs within 1 month prior to Screening Visit
* Thyroid hormones or preparations within 1 month prior to Screening Visit (except in subjects on stable dose of replacement therapy for at least 1 month)
* Thiazide diuretics within 2 weeks prior to Screening Visit
* Discontinuation of beta-blockers within 1 month prior to Screening Visit or planned discontinuation of beta-blocker therapy
* Anticipated requirement for use of prohibited concomitant medications

History of allergic reaction or significant intolerance to:

* Diazoxide
* Thiazides
* Sulfonamides
* Fenofibrate or fenofibric acid derivatives

Lifestyle changes

• Subjects intending to change exercise habits, quit smoking and/or quit alcohol use during the entire study

Specific diagnoses, medical conditions and history

* Known type I or III hyperlipidemia
* Known type 1 DM
* Current diagnosis of type 2 DM
* Any other clinically significant endocrine, cardiovascular, pulmonary, neurological, psychiatric, hepatic, gastrointestinal, hematological, renal, or dermatological disease interfering with the assessments of the study medications, according to the Investigator

Specific laboratory test results

• Any relevant biochemical abnormality interfering with the assessments of the study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Triglyceride-lowering efficacy of DCCR | 84 days
  Fasting triglycerides (percent change from Baseline to Day 84)

SECONDARY OUTCOMES:
Improvement in other lipid profiles with DCCR | 84 days
  Apolipoprotein B (Apo B) (percent change from Baseline to Day 84) Fasting non-HDL cholesterol (percent change from Baseline to Day 84)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Baron, M.D., Study Director — Essentialis, Inc.